CLINICAL TRIAL: NCT05245357
Title: Therapeutic Impacts of Dietary Pulses on Bile Acids
Brief Title: Impact of Foods on Bile Acids, Metabolites, and Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Montana State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AFRI Grant 2021-67028-34103
Record Dates: First submitted 2022-01-31; First posted 2022-02-17 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Inflammation; Hypertriglyceridemia; Metabolic Disease; Lipid Metabolism Disorder; Hyperlipidemias; Bile Acid Malabsorption
MeSH Terms: conditions — Inflammation; Hypertriglyceridemia; Metabolic Diseases; Lipid Metabolism Disorders; Hyperlipidemias | interventions — lentil lectin

STUDY DESIGN:
Intervention Model Description: The design is 2 x 2 crossover design, where the overweight and obese adults without Type 2 Diabetes will be randomized into Control or Lentil
Who Masked: Participant, Investigator
Masking Description: Lentil and Control meals were designed to be comparable in taste and appearance. The meals are prepared and coded prior to receipt by the research team. Randomization is for order of coded meals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lentil, then Control (Experimental): Participants first received a meal with 140 g of lentils in the morning. After a washout period of at least 7 days, they then received a meal with 0 g of lentils in the morning.
  Interventions: Behavioral: Lentil; Behavioral: Control
- Control, then Lentil (Experimental): Participants first received a meal with 0 g of lentils in the morning. After a washout period of at least 7 days, they then received a meal with 140 g of lentils in the morning.
  Interventions: Behavioral: Lentil; Behavioral: Control

INTERVENTIONS:
Behavioral: Lentil — Participants in the lentil arm of the study will consume a meal containing 140 g of lentils for breakfast one morning.
Behavioral: Control — Participants in the control arm of the study will consume a meal containing 0 g of lentils for breakfast one morning.

SUMMARY:
Dietary incorporation of pulse crops may be an effective way to lower unhealthy elevations in serum bile acids. These elevations play a direct role in promoting obesity-related diseases estimated to be present in about one third of the US adult population, including non-alcoholic fatty liver disease and type 2 diabetes. The overarching hypothesis for this study is that pulse consumption increases bile acid secretion and excretion, which will decrease toxicity linked to excess accumulation of bile in the liver, improve metabolism, and lower resulting levels of bile acids in the serum. In direct alignment with the USDA-AFRI Food, Safety, Nutrition, and Health priority to address obesity and related chronic disease with increased fruit and vegetable consumption and also with the American Pulse Association call to investigate the impact of regular pulse consumption on human physical well- being, the long-term research goal of this study is to establish effective and practical therapeutic strategies utilizing dietary incorporation of pulse crops to prevent or reverse obesity driven diseases. The specific objectives in this proposal are to:

1. determine the impact of acute lentil ingestion on serum postprandial bile acid responses and composition in a human cohort with obesity, and
2. determine the impact of daily lentil consumption for 12 weeks on serum fasting and postprandial bile acid concentrations and composition in an overweight or obese cohort with elevated postprandial triglycerides.

This proposal is being submitted in response to the American Pulse Association commodity board sponsored topic of investigating the impact pulse crop consumption on health.

DETAILED DESCRIPTION:
The approach for Objective 1 is to enroll a population of overweight/obese individuals (n=24) in a two-armed (LENTIL and CONTROL), randomized, crossover trial in which each individual participant serves as his/her own control to compare postprandial serum bile acid responses between isocaloric meals with the same amount of fat with (LENTIL) and without (CONTROL) lentils. Isocaloric meals with the same total fat content in LENTIL and CONTROL study arms will provide the same stimulus to induce increased postprandial serum bile acids. The randomized crossover design with half of the participants starting in the LENTIL arm and the other half starting in the CONTROL arm will eliminate potential order effects. Block randomization with 3 blocks of two equally numbered levels (total of 8 per block) will be created. Having each person serve as their own control in a crossover trial will eliminate the influence of inter-individual variation. The MSU Nutrition Research team has extensive experience with postprandial testing protocols and dietary manipulation and will utilize this experience to perform the proposed protocol with appropriate pre-test standardization, uniformity of meal preparation, precise timing of blood collection, and established procedures for processing and analyzing blood samples. Bile acids, including all primary and secondary forms, will be analyzed from samples collected before the meal and at 30-minute intervals for 4 hours after the meal. Established methods in the MSU Proteomics, Metabolomics, and Mass Spectrometry Facility will be used to compare total and individual bile acids between LENTIL and CONTROL conditions.

The approach for Objective 2 will leverage banked samples from a highly synergistic ongoing clinical trial comparing 12 weeks of daily lentil consumption to control. This study utilizes a randomized, parallel research design to compare the impact of ingesting 140 g of lentils per day to 0 g per day for 12 weeks on serum triglyceride and inflammation responses to a high-fat meal. High fat meals induce the largest serum bile acid responses so the current proposal augments this study by adding assessment of the impact of prolonged lentil consumption on the appearance of bile acids in the systemic circulation under fasting and postprandial conditions. In contrast to Objective 1, which focuses on the acute impact of incorporating lentils into a meal, Objective 2 will measure the impact of adaptations to lentil ingestion that improve enterohepatic function. These changes may be facilitated by changes to the composition of the gut microbiome, enhanced bile acid excretion, or other mechanisms independent of having lentils in the challenge meal. Data from the ongoing trial will be analyzed to determine whether lentils induced changes in the composition of the gut microbiome. This proposal will analyze whether lentil consumption increases excretion of bile acids by analyzing bile acid composition of stool samples collected before and after lentil supplementation. In sum, adding analysis of serum and stool bile acids from samples collected and banked in an ongoing clinical trial, will allow the determination of whether lentil consumption over time improves enterohepatic health in a way that reduces appearance of bile acids in serum and or increases excretion of bile acids.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years of age
* Body Mass Index greater than 27 kg/m^2

Exclusion Criteria:

* taking medication that will influence cholesterol, lipids, or inflammation
* a gallbladder condition or have had the gallbladder removed
* allergy to wheat, dairy, or legumes
* pregnant or lactating
* have been on a ketogenic or paleo diet in the past 6 weeks
* have been on antibiotics in the past 90 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Postprandial Bile Acid Response to High-Fat Meal | 1 day
  Area under the curve for bile acid concentration after consuming a meal containing 40g fat
Peak Bile Acid Response to High-Fat Meal | 1 day
  Greatest change in bile acid concentration after consuming a meal containing 40g fat
Postprandial Triglyceride Response to High-Fat Meal | 1 day
  Area under the curve for triglcyerides concentration after consuming a meal containing 40g fat
Peak Triglyceride Response to High-Fat Meal | 1 day
  Greatest change in triglycerides concentration after consuming a meal containing 40g fat
Postprandial Serum Inflammatory Cytokine (tumor necrosis factor-alpha, interleukin-(IL)1beta, IL-6, IL-10, IL-17, IL-23, interferon-gamma, and granulocyte macrophage-colony stimulating factor; all in pg/ml) Response to High-fat Meal | 1 day
  Area under the curve for inflammatory cytokine (tumor necrosis factor-alpha, interleukin-(IL)1beta, IL-6, IL-10, IL-17, IL-23, interferon-gamma, and granulocyte macrophage-colony stimulating factor; all in pg/ml) concentrations after consuming a meal containing 40 g of fat
Postprandial Serum Metabolite Response (untargeted) to a High-Fat Meal | 1 day
  Changes in concentrations of metabolites measured with untargeted liquid chromatography mass spectrometry (LCMS) metabolomic analysis after consuming a meal containing 40g of fat
Fasting Serum Metabolite Response (untargeted) to a High-Fat Meal | 1 day
  Changes in concentrations of metabolites measured with untargeted liquid chromatography mass spectrometry (LCMS) metabolomic analysis before consuming a meal containing 40g of fat
Gut Microbiome Composition | 1 day
  Relative abundance of operational taxonomic units of microbes measured from fecal samples

SECONDARY OUTCOMES:
Body Composition | 1 day
  % body fat
Visceral Adipose Tissue | 1 day
  Quantity of adipose in liters located within the abdominal compartment
Body Mass Index | 1 day
  kg of body mass per meter of height squared
Habitual Diet | 1 month
  Habitual dietary intake from past month reported through a food frequency questionnaire for food, beverage, and supplement intake
Acute Diet | 1 day
  Dietary intake from the last 24-hours, self-reported through a guided online prompt
Acute Physical Activity | 1 day
  Physical activities from the last 24-hours, self-reported through a guided online promoted

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Miles, PhD, Principal Investigator — Montana State University
Locations (1):
- Nutrition Research Laboratory, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No